CLINICAL TRIAL: NCT00754559
Title: "Effectiveness After Four and Twentyfour Weeks and Safety of Tocilizumab in Patients With Active RA"
Brief Title: A Study to Assess Efficacy With Respect to Clinical Improvement in Disease Activity and Safety of Tocilizumab in Patients Wtih Active Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21469; 2008-000105-11
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 8mg/kg iv every 4 weeks

SUMMARY:
This single arm study will assess the effectiveness of tocilizumab in combination with traditional DMARDs with regard to the clinical improvement in disease activity (achievement of LDAS) after 24 weeks' treatment in patients with active rheumatoid arthritis (RA) who have had an inadequate response to current traditional DMARD and/or anti-TNF therapy. Patients will receive tocilizumab 8mg/kg iv every 4 weeks, in addition to ongoing DMARDs at the stable pre-entry dose prescribed by the physician, for a total of 6 infusions during the regular treatment period and a further 6 infusions during an optional extension phase. The anticipated time on study treatment is 6 to 12 months, and the target sample size is <500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* rheumatoid arthritis of >=6 months duration diagnosed according to the revised 1987 ACR criteria;
* DAS28 of >3.2;
* At screening either ESR >=28 mm/h or CRP >=1 mg/dL;
* Having received permitted DMARDs, 1 or more; current DMARD therapy must have been at a stable dose for at least 8 weeks prior to baseline.

Exclusion Criteria:

* major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following screening;
* functional class IV as identified by the ACR classification of functional status in RA;
* rheumatoid autoimmune disease other than RA;
* prior history of or current inflammatory joint disease other than RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2008-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- Germany (61):
  - Aachen
  - Bad Abbach
  - Bad Aibling
  - Bad Bramstedt
  - Bad Nauheim
  - Baden-Baden
  - Bayreuth
  - Berlin
  - Bremen
  - Cologne
  - Cuxhaven
  - Damp
  - Donaueschingen
  - Dresden
  - Düsseldorf
  - Erfurt
  - Erlangen
  - Essen
  - Frankfurt
  - Frankfurt am Main
  - Fulda
  - Gommern
  - Goslar
  - Göttingen
  - Grafschaft
  - Hagen
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Hildesheim
  - Hofheim
  - Homburg/saar
  - Hoyerswerda
  - Leipzig
  - Ludwigsfelde
  - Ludwigshafen
  - Lüneburg
  - Mainz
  - Marburg
  - München
  - Münster
  - Naunhof
  - Neuss
  - Nuremberg
  - Oberammergau
  - Osnabrück
  - Pirna
  - Plochingen
  - Potsdam
  - Ratingen
  - Rostock
  - Sendenhorst
  - Stuttgart
  - Treuenbrietzen
  - Tübingen
  - Ulm
  - Wiesbaden
  - Würselen
  - Zeven

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams/kilogram (mg/kg) intravenously (iv) every 4 weeks for a total of 6 infusions.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 286
Completed | 239
Not Completed | 47
Not completed — Adverse Event | 15
Not completed — Protocol Violation | 11
Not completed — Lack of Efficacy | 10
Not completed — Lost to Follow-up | 2
Not completed — Administrative reason | 1
Not completed — Other | 5
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All treated participants were included in the safety population as well as the intent to-treat (ITT) population.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg iv every 4 weeks for a total of 6 infusions.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Low Disease Activity Score at Week 24
Description: Low Disease Activity Score (LDAS) is defined as Disease Activity score less than or equal to (≤ ) 3.2. Disease activity score 28 (DAS28) was calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and global health assessment (participant rated global assessment of disease activity using 100-mm Visual analog scale [VAS]); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity.
Time Frame: Week 24
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
Percentage of Participants | 57 [51 to 62.8]
Statistical Analysis 1: Comparison: Tocilizumab; Null hypothesis: Proportion of participants reaching LDAS (≤ 3.2) at Week 24 equals (=) expected proportion of 42%; Test type: Superiority or Other; p < 0.001, Exact Binomial Test

2. Secondary Outcome: Absolute Changes in DAS28 From Baseline
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant rated global assessment of disease activity using 100-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 ≤3.2 = low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population; only participants with a DAS28 value at baseline were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 274
units on a scale
  Week 1 | -1.31 (1.1)
  Week 2 | -2.1 (1.2)
  Week 4 | -2.4 (1.2)
  Week 8 | -2.8 (1.3)
  Week 12 | -3.2 (1.4)
  Week 16 | -3.2 (1.4)
  Week 20 | -3.3 (1.4)
  Week 24 | -3.4 (1.4)

3. Secondary Outcome: Percentage of Participants With a Response at Week 24 by European League Against Rheumatism (EULAR) Category
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 ≤3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or change from baseline >0.6 to ≤1.2 with DAS28 ≤5.1; non-responders: change from baseline ≤ 0.6 or change from baseline >0.6 and ≤1.2 with DAS28 >5.1.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
Percentage of Participants
  Good | 54.9
  Moderate | 20.3
  None | 24.8

4. Secondary Outcome: Percentage of Participants With a DAS28 Response at Weeks 4 and 24
Description: DAS28 calculated from the number of swollen joints and painful joints using the 28-joint count, the ESR and participant's global assessment (PGA) of disease activity (participant rated arthritis activity assessment using VAS) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 ≤3.2 = low disease activity, DAS28 <2.6 = remission and a clinically significant (CS) reduction was defined as ≥1.2.
Time Frame: Weeks 4 and 24
Population: ITT Population;
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
percentage of participants
  Week 4, CS reduction | 75.2 [69.7 to 80.1]
  Week 4, Remission | 23.1 [18.3 to 28.4]
  Week 4, CS reduction or remission | 76.6 [71.2 to 81.4]
  Week 4, LDAS | 40.9 [35.2 to 46.9]
  Week 24, CS reduction | 74.5 [69.0 to 79.4]
  Week 24, Remission | 47.6 [41.6 to 53.5]
  Week 24, CS reduction or remission | 76.6 [71.2 to 81.4]
  Week 24, LDAS | 57.0 [51.0 to 62.8]

5. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20%, 50%, or 70% (ACR20/ACR50/ACR70) Response
Description: ACR20/50/70 response: ≥20%, 50%, or 70% improvement, respectively, in swollen and tender joint count; and ≥20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ-DI]); and C-Reactive Protein (CRP).
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
percentage of participants
  Week 1 ACR20 | 25.2 [20.3 to 30.6]
  Week 1 ACR50 | 7.0 [4.3 to 10.6]
  Week 1 ACR70 | 2.4 [1.0 to 5.0]
  Week 2 ACR20 | 41.3 [35.5 to 47.2]
  Week 2 ACR50 | 14.7 [10.8 to 19.3]
  Week 2 ACR70 | 4.9 [2.7 to 8.1]
  Week 4 ACR20 | 50.0 [44.1 to 55.9]
  Week 4 ACR50 | 25.5 [20.6 to 31.0]
  Week 4 ACR70 | 12.2 [8.7 to 16.6]
  Week 8 ACR20 | 64.3 [58.5 to 69.9]
  Week 8 ACR50 | 37.4 [31.8 to 43.3]
  Week 8 ACR70 | 17.1 [13.0 to 22.0]
  Week 12 ACR20 | 69.6 [63.9 to 74.9]
  Week 12 ACR50 | 48.6 [42.7 to 54.6]
  Week 12 ACR70 | 26.2 [21.2 to 31.7]
  Week 16 ACR20 | 67.5 [61.7 to 72.9]
  Week 16 ACR50 | 49.0 [43.0 to 54.9]
  Week 16 ACR70 | 29.4 [24.2 to 35.0]
  Week 20 ACR20 | 67.8 [62.1 to 73.2]
  Week 20 ACR50 | 49.7 [43.7 to 55.6]
  Week 20 ACR70 | 33.9 [28.4 to 39.7]
  Week 24 ACR20 | 65.0 [59.2 to 70.6]
  Week 24 ACR50 | 50.7 [44.7 to 56.6]
  Week 24 ACR70 | 33.9 [28.4 to 39.7]

6. Secondary Outcome: Change From Baseline in Swollen and Tender Joint Counts at Week 24
Description: Swollen joint count: 66 joints were assessed for swelling and joints were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
  Tender joint counts: 68 joints were assessed for tenderness and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
Time Frame: Week 24
Population: ITT Population; missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (95% Confidence Interval); unit: Joints
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg iv every 4 weeks up to week 20 for a total of 6 infusions.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
Joints
  Number of swollen joints | -9.6 [-10.4 to -8.7]
  Number of tender joints | -13.4 [-14.7 to -12.1]

7. Secondary Outcome: Change From Baseline in the Levels of C-Reactive Protein at Week 24
Description: The serum concentration of CRP is measured in mg/L. A reduction in the level was considered an improvement.
Time Frame: Week 24
Population: ITT Population; missing data were imputed using LOCF.
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mg/L | -20.1 [-23.7 to -16.6]

8. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Pain (VAS) at Week 24
Description: Participant's global assessment of pain was assessed using a 100-mm horizontal VAS (0 to 100 mm) with 0=pain absent and 100=unbearable pain. Participants responded by placing a mark on the line to indicate their current level of pain.
Time Frame: Week 24
Population: ITT Population; missing data were imputed using LOCF.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mm | -36.2 [-39.6 to -32.7]

9. Secondary Outcome: Change From Baseline in Participant and Physician Assessment of Global Disease Activity (VAS) at Week 24
Description: Participant's global assessment of disease activity was an overall assessment of their current disease activity on a 100-mm horizontal VAS scale (left-hand extreme: "no disease activity"; right-hand extreme: "maximum disease activity").
  Physician's global assessment of disease activity was measured as participant's current disease activity on a 100-mm horizontal VAS scale (left hand extreme: "no disease activity"; right-hand extreme: "maximum disease activity").
Time Frame: Week 24
Population: ITT Population; missing data were imputed using LOCF.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mm
  Participant's assessment | -35.9 [-39.5 to -32.4]
  Physician's assessment | -44.9 [-47.7 to -42.1]

10. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score
Description: CDAI was calculated according to the following formula:
  CDAI = Number of swollen joints (plus) + Number of tender joints + VAS disease activity participant assessment + VAS disease activity investigator assessment. The maximum score was 334 (66 joints + 68 joints + 100 mm + 100 mm); higher scores indicated higher disease activity.
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population; only participants with values for CDAI at baseline and the respective visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
units on a scale
  Week 1 | -8.4 (12.1)
  Week 2 | -13.3 (12.4)
  Week 4 | -15.6 (13.4)
  Week 8 | -19.7 (13.2)
  Week 12 | -22.4 (13.4)
  Week 16 | -22.4 (13.8)
  Week 20 | -22.7 (13.3)
  Week 24 | -24.2 (12.9)

11. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Week 24
Population: ITT Population; Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
units on a scale | -0.48 (0.60)

12. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 24
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status.
Time Frame: Week 24
Population: ITT Population; Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
units on a scale | 8.6 (11.1)

13. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Score at Week 24
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Absolute change was defined as the change from baseline to Week 24.
Time Frame: Week 24
Population: ITT Population; Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tocilizumab: Participants received tocilizumab 8mg/kg iv every 4 weeks up to week 20 for a total of 6 infusions.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
units on a scale
  Physical functioning | 18.4 (24.6)
  Role physical | 16.5 (21.6)
  Bodily pain | 25.0 (22.3)
  General health perception | 11.9 (18.7)
  Vitality | 18.0 (20.2)
  Social functioning | 13.8 (27.2)
  Role emotional | 13.9 (50.1)
  Mental health | 10.3 (19.1)

14. Secondary Outcome: Participant's Global Assessment of Pain as Assessed by Patient Take Home Form (PTHF)
Description: Participant's were asked to state the worst level of pain felt in the past 24 hours using a 100-mm horizontal VAS (0 to 100 mm) with 0=no pain and 100=unbearable pain. Participants responded by placing a mark on the line to indicate their level of pain. Participants were asked to document their response during the first 4 treatment weeks at approximately the same time every day.
Time Frame: Baseline and Weeks 1, 2, and 4
Population: ITT Population; Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mm
  Baseline | 60.7 (23.1)
  Week 1 | 48.6 (25.2)
  Week 2 | 41.9 (25.4)
  Week 4 | 36.3 (26.7)
  Change at Week 1 | -12.0 (22.3)
  Change at Week 2 | -18.7 (24.9)
  Change at Week 4 | -24.4 (27.4)

15. Secondary Outcome: Duration of Morning Stiffness as Assessed Using PTHF
Description: Duration of morning stiffness: participants were asked 'how long did your morning stiffness last from the time you woke up yesterday' and the response was provided in minutes and hours. Participants were asked to document their response during the first 4 treatment weeks at approximately the same time every day.
Time Frame: Baseline, Weeks 1, 2, and 4
Population: ITT Population; Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
hours
  Baseline | 2.4 (2.8)
  Week 1 | 1.8 (2.3)
  Week 2 | 1.5 (1.8)
  Week 4 | 1.2 (1.5)
  Change at Week 1 | -0.6 (1.8)
  Change at Week 2 | -0.9 (2.1)
  Change at Week 4 | -1.2 (2.3)

16. Secondary Outcome: Participant Assessment of Fatigue/Tiredness as Assessed Using PTHF
Description: Participants were asked to assess their overall level of fatigue/tiredness during the previous 24 hours using a 100-mm horizontal VAS with 0=none and 100=very severe. Participants responded by placing a mark on the line to indicate their current level of fatigue. Participants were asked to document their response during the first 4 treatment weeks at approximately the same time every day.
Time Frame: Baseline and Weeks 1, 2 and 4
Population: ITT Population; Missing data were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mm
  Baseline | 52.9 (26.9)
  Week 1 | 42.2 (26.2)
  Week 2 | 36.3 (26.5)
  Week 4 | 30.6 (26.0)
  Change at Week 1 | -10.6 (22.0)
  Change at Week 2 | -16.6 (24.1)
  Change at Week 4 | -22.2 (26.5)

17. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Score
Description: The TSQM is a general measure of participants treatment satisfaction and consists of 14 questions that result in 4 subscales: "effectiveness", "side-effects", "convenience" and "global satisfaction". All subscale scores range from 0 to 100%, with 100% being the best possible result.
Time Frame: Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
units on a scale
  Percent Effectiveness | 69.4 (28.3)
  Percent Side-effects | 88.7 (21.7)
  Percent Convenience | 72.4 (20.8)
  Percent Global satisfaction | 74.7 (25.9)

18. Secondary Outcome: Changes in Hemoglobin
Description: Hemoglobin levels were determined as a hematology parameter to measure changes in disease related anemia.
Time Frame: Baseline, Weeks 1, 2, 4 and 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
g/dL
  Baseline | 128.6 (13.1)
  Week 1 | 132.2 (13.4)
  Week 2 | 133.5 (13.1)
  Week 4 | 133.5 (13.6)
  Week 24 | 136.1 (13.7)
  Change at Week 1 | 3.5 (6.8)
  Change at Week 2 | 4.8 (6.5)
  Change at Week 4 | 4.3 (8.0)
  Change at Week 24 | 7.5 (9.7)

19. Secondary Outcome: Changes in C-Reactive Protein
Description: CRP is an acute phase inflammatory marker used as a measure of inflammation. A reduction in CRP is considered to be an improvement.
Time Frame: Baseline, Weeks 1, 2 ,4 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mg/L
  Baseline | 23.1 (30.7)
  Week 1 | 3.5 (6.6)
  Week 2 | 2.4 (4.4)
  Week 4 | 5.5 (14.8)
  Week 24 | 3.0 (7.7)
  Change at Week 1 | -19.6 (29.4)
  Change at Week 2 | -20.7 (29.8)
  Change at Week 4 | -17.5 (27.7)
  Change at Week 24 | -20.1 (29.9)

20. Secondary Outcome: Changes in Erythrocyte Sedimentation Rate (ESR)
Description: ESR is an inflammation marker used to determine acute phase response.
Time Frame: Baseline, Weeks 1, 2, 4 and 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Tocilizumab
Number analyzed (Participants) | 286
mm/h
  Baseline | 37.4 (22.1)
  Week 1 | 16.7 (14.2)
  Week 2 | 10.6 (11.0)
  Week 4 | 10.3 (13.5)
  Week 24 | 7.1 (9.5)
  Change at Week 1 | -20.6 (17.9)
  Change at Week 2 | -26.7 (19.0)
  Change at Week 4 | -27.2 (18.6)
  Change at Week 24 | -30.3 (21.7)

21. Secondary Outcome: Percentage of Participants Withdrawing From Study Treatment Because of Insufficient Therapeutic Response
Description: Participants who withdrew from study drug due to other reasons were not taken into account.
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population; participants who withdrew from study drug due to other reaasons were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tocilizumab: Participants received tocilizumab 8mg /kg iv every 4 weeks for a total of 6 infusions.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 249
percentage of participants | 4.0 [1.9 to 7.3]

ADVERSE EVENTS:
Time Frame: Adverse events were reported throughout the study including any reactions that occurred within 24 hours after infusion.
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 32/286
Other Adverse Events (participants affected / at risk) | 242/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=286)
Pneumonia (Infections and infestations) | 2
Abscess jaw (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pharyngeal abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Low density lipoprotein increased (Investigations) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
General physical health deterioration (General disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Chest pain (General disorders) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 8
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=286)
Eosinophilia (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 2
Intravascular haemolysis (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Extrasystoles (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachyarrhythmia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 4
Cushingoid (Endocrine disorders) | 1
Goitre (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 6
Dry eye (Eye disorders) | 1
Eye inflammation (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 4
Aphthous stomatitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 16
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Enteritis (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Gingival erythema (Gastrointestinal disorders) | 1
Loose tooth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Periodontitis (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Discomfort (General disorders) | 3
Drug intolerance (General disorders) | 3
Fatigue (General disorders) | 13
General physical health deterioration (General disorders) | 1
Local swelling (General disorders) | 1
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 6
Pitting oedema (General disorders) | 1
Thirst (General disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Food allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 5
Seasonal allergy (Immune system disorders) | 2
Abscess jaw (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 16
Bronchopneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 5
Eyelid infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 3
Fungal skin infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Gastrointestinal infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Herpes zoster ophthalmic (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Lower respiratory tract infection viral (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 54
Onychomycosis (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 6
Osteomyelitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 3
Paronychia (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pharyngeal abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Post procedural infection (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Prostate infection (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 15
Septic shock (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 8
Skin bacterial infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 9
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 15
Urinary tract infection bacterial (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 4
Vulvitis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Nail injury (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 8
Radius fracture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 24
Aspartate aminotransferase increased (Investigations) | 14
Basophil count increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 4
Blood cholesterol increased (Investigations) | 5
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 2
Blood uric acid increased (Investigations) | 2
Body temperature increased (Investigations) | 2
Haematocrit increased (Investigations) | 1
Haemoglobin increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 79
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Transaminases increased (Investigations) | 2
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 6
Hyperureicaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Facit joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 25
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dysaesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Facial neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 27
Migraine (Nervous system disorders) | 4
Multiple sclerosis relapse (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Synope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 2
Food aversion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Mood altered (Psychiatric disorders) | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 3
Haematuria (Renal and urinary disorders) | 3
Leukocyturia (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Breast disorder (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Genital cyst (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 2
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin chapped (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 16
Lymphoedema (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights